CLINICAL TRIAL: NCT04526067
Title: In-person vs. Remote Wellness Support (Study Sub-title: Remote Cognitive Adaptation Training to Improve Medication Follow Through in Managed Care (R-CAT))
Brief Title: In-person vs. Remote Wellness Support
Acronym: R-CAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20200525H; 1R56MH123797 (NIH)
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Depressive Disorder, Major; Bipolar Disorder; Schizo Affective Disorder; Schizophrenia
Keywords: Serious mental illness
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Intervention Model Description: Randomized parallel design
Who Masked: Outcomes Assessor
Masking Description: Those with no preference for CAT or R-CAT will be Randomized, 1:1 done by statistician who has no patient contact through a random allocation program. If blinds are broken accidentally, new raters can be assigned, but blinds are kept by having raters and pill counters unaware of treatment group or study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Adaptation Training (CAT) (Active Comparator): A home delivered adherence intervention used by managed care used to improve outcomes across multiple conditions.
  Interventions: Behavioral: CAT
- Remote Cognitive Adaptation Training (R-CAT) (Active Comparator): A primarily remotely delivered workable adherence intervention used by managed care used to improve outcomes across multiple conditions.
  Interventions: Behavioral: R-CAT

INTERVENTIONS:
Behavioral: CAT — An evidence-based psychosocial treatment using environmental supports such as signs, alarms, pill containers, and the organization of belongings established in a person's home on weekly visits to cue adaptive behaviors and establish healthy habits.
  Other Names: Cognitive Adaptation Training
  Arms: Cognitive Adaptation Training (CAT)
Behavioral: R-CAT — An evidence-based psychosocial treatment using environmental supports such as signs, alarms, pill containers, and the organization of belongings established in a person's home using remote weekly visits to cue adaptive behaviors and establish healthy habits.
  Other Names: Remote Cognitive Adaptation Training
  Arms: Remote Cognitive Adaptation Training (R-CAT)

SUMMARY:
The study team will use components of the Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) framework to compare Cognitive Adaptation Training (CAT) to Remotely delivered Cognitive Adaptation Training (R-CAT) 1-9 within a managed care organization (MCO), targeting members with serious mental illness (SMI) needing assistance with the regular taking of medication.

DETAILED DESCRIPTION:
Individuals choosing or assigned to R-CAT will continue treatment as usual with their health care team and R-CAT will be added. R-CAT is a remotely delivered version of CAT focused on medication adherence using a series of manual-driven compensatory strategies and environmental supports (signs, checklists, electronic cueing devices) based upon a streamlined assessment of executive function impairment and barriers to habit formation including forgetfulness, difficulties in problem-solving, disorganization, apathy or amotivation, disinhibition. and home environment. Initial R-CAT goals are to 1) ensure that medications listed as prescribed are available 2) to assess current cognitive, behavioral and environmental facilitators and barriers to habit-formation 3) to set up customized CAT supports to address the barriers and use facilitators to build habits to take medication. Rare home visits may occur if issues cannot be resolved remotely. Based upon the pilot, the study team don't anticipate any more than 5-10% of individuals to need face-to-face visits. No one had home visits as part of the pilot intervention. A structured R-CAT treatment note with places for pictures of CAT interventions is used for home visits. Support and reminder calls use a brief checklist modified from the Healthy Habits Program to address issues in use of supports, placement of supports and habit formation. Examples of CAT interventions to promote taking medication regularly appear above. All home visits and phone calls will be audio-taped (with consent) for quality assurance.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give informed consent.
2. Between the ages of 18 and 65.
3. Clinical Diagnosis of Major Depressive Disorder, Bipolar disorder, Schizophrenia, or Schizoaffective Disorder
4. Receiving treatment with oral psychiatric medications.
5. Have had a hospitalization or emergency department visit in the past year
6. Have a Medication Possession Ratio (MPR) based upon electronic refill data below 80% at least 1 of the past 4 quarters with at least 1 psychiatric medication
7. Responsible for taking their own medications
8. Report on telephone prescreen call with researcher team that they have missed at least 2 doses of medication in the past 3 weeks, that they are willing to take medication and would like remote assistance to take medication more regularly
9. Report on telephone prescreen call with research team that they have a stable living environment (individual apartment, family home, board and care facility) within the last three months and no plans to move in the next year
10. Report on prescreen research call with research team that they have no plans to change their MCO in the next 12 months
11. Have a working smart phone
12. Able to understand and complete rating scales and assessments.
13. Agree to home visits for intervention and to count pills and conduct assessments

Exclusion Criteria:

1. Substance dependence within the past 2 months
2. Currently being treated by an ACT team
3. Documented history of violence or threatening behavior on initial assessment
4. Receive home visits to assist with medication adherence
5. Unable to complete baseline assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Velligan, PhD, Principal Investigator — University of Texas Health at San Antonio
Locations (1):
- University of Texas Health Science Center - Department of Psychiatry, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Because this is a research study, we will be unable keep your PHI completely confidential. We may share your health information with people and groups involved in overseeing this research study including:
  * The National Institute of Mental Health who is funding this study
  * The following collaborators at other institutions that are involved with the study: Superior Medicaid
  * The committee that checks the study data on an ongoing basis, to determine if the study should be stopped for any reason.
  * The members of the local research team
  * The Institutional Review Board and the Compliance Office of the University of Texas Health Science Center at San Antonio, and other groups that oversee how research studies are carried out.
Supporting Information: Study Protocol, SAP
Time Frame: Data may be shared with individuals or groups overseeing this project for reporting purposes throughout the study life and after study completion, unidentified participant data will be shared at the time of publication.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were 56 members of a large Managed Medicaid program in Texas
Groups:
- R-CAT: While the original design called for participants to either be randomized to CAT or R-CAT or to indicate a preference and be assigned to these groups, due to risk of COVID-19 infection during the pandemic, only R-CAT could be offered during the early parts of the trial. Therefore, 21 individuals were simply assigned to R-CAT and 14 received R-CAT based upon preference. This treatment group provided Cognitive Adaptation Remotely via secure video conference, sent text message reminders, delivered environmental supports by mail. Environmental supports targeted medication and appointment follow-through, independent living skills and organization, and socialization. Supports were set up on virtual visits conducted weekly.
- CAT Cognitive Adaptation Training: While the original design called for participants to either be randomized to CAT or R-CAT or to indicate a preference and be assigned to these groups, due to risk of COVID-19 infection during the pandemic, only R-CAT could be offered during the early parts of the trial. 21 participants received CAT based upon preference for CAT versus R-CAT. CAT involved in person assessment and establishing supports in the home for medication follow-through, independent living skills/organization and socialization.
Period: Overall Study
Arm/Group | R-CAT | CAT Cognitive Adaptation Training
Started (Completers had baseline and at least one follow-up assessment) | 35 | 21
Completed (Completers had baseline and at least one follow up assessment) | 35 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Adaptation Training (CAT) | Remote Cognitive Adaptation Training (R-CAT) | Total
Number analyzed (Participants) | 21 | 35 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (14.0) | 44.8 (10.7) | 44.9 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 13 | 26 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 12 | 13
  White | 19 | 19 | 38
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 1 | 2
Social and Occupational Functioning Scale score [Mean (Standard Deviation); unit: units on a scale] — The Social and Occupational Functioning Assessment Scale (SOFAS) is a rating scale that measures a patient's current functioning on a scale of 0 to 100, with lower scores indicating lower functioning. The SOFAS is based on a clinician's judgment of a patient's functioning in four areas: Socially useful activities, Personal and social relationships, Self-care, and Disturbing and aggressive behaviors.
  units on a scale | 39.1 (2.4) | 44.9 (1.9) | 42.72 (2.09)

OUTCOME MEASURES:

1. Primary Outcome: Acceptance of Intervention-Number of Participants Who Dropped Out of Treatment
Description: Proportion of subjects who dropped out of treatment
Time Frame: Baseline to 6 months
Population: examined descriptive statistics for proportion of drop outs by group
Measure: Count of Participants; unit: Participants
Arm/Group | R-CAT | CAT Cognitive Adaptation Training
Number analyzed (Participants) | 35 | 21
Participants | 4 | 3

2. Primary Outcome: Medication Adherence
Description: Adherence proportion is calculated as the number of pills missing and presumed taken/ the number of pills prescribed for the time period. Monthly checks will be performed.
Time Frame: Baseline to 6 months
Population: IIT population with baseline and at least 1 follow up
Measure: Mean (Standard Error); unit: proportion of pills taken
Arm/Group | R-CAT | CAT Cognitive Adaptation Training
Number analyzed (Participants) | 35 | 21
proportion of pills taken | .21 (0.05) | .10 (0.08)

3. Primary Outcome: Functional Outcome
Description: Functional outcome will be rated using the Social and Occupational Functioning Scale (SOFAS).The SOFAS rates functioning on a scale from 0 to 100 based upon all the data collected in the assessment. Higher scores reflect better functional outcome. The value reported is the the 6 month value minus the baseline value>
Time Frame: Baseline to 6 months note that repeated measures analysis was also used
Population: ITT population with at least a baseline and one follow-up assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | R-CAT | CAT Cognitive Adaptation Training
Number analyzed (Participants) | 35 | 21
score on a scale | 1.88 (1.72) | 6.48 (2.08)

4. Secondary Outcome: Self-Report Habit Index (SRHI)
Description: A 36-item scale assessing three types of habit taking medication, following a schedule or calendar, and grooming (specifically brushing teeth. 12 items assessed each behavior; The SRHI looks at 1) automaticity , 2) frequency, and 3) relevance to self-identity for each behavior.
  There are 12 items for each sub-scale scored 1-7 (total possible range is 12-84 for each of the 3 scales). A total Habit score will be computed by calculating the mean of the 3 sub-scales to give a value between 12 and 84. Lower mean scores indicate greater habit strength.
Time Frame: Baseline to 6 months (note that repeated measures analysis examined change over time as well.
Population: IIT analysis of all with baseline and at least 1 follow up assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | R-CAT | CAT Cognitive Adaptation Training
Number analyzed (Participants) | 35 | 21
score on a scale | 6.6 (2.69) | 7.6 (3.27)

5. Secondary Outcome: Symptomatology
Description: Change in symptoms assess by a trained rater using the Brief Psychiatric Rating Scale-Expanded Version (BPRS-E). The scale is used to rate the subjects using 24 items, each to be rated in a 7-point scale of severity ranging from NA (not assessed), then 1-7, with 7 being the most severe. The possible range of scores is from 1 to 168 with a total score reflects an overall level of symptomology, with 168, being the maximum score, with the most symptoms present. The value reported is the 6 month value minus the baseline value.
Time Frame: Baseline to 6 months
Population: ITT sample with baseline and at least one follow up. Also conducted repeated measures analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Remote Cognitive Adaptation Training (R-CAT) | Cognitive Adaptation Training (CAT)
Number analyzed (Participants) | 35 | 21
score on a scale | 13.7 (2.5) | 6.82 (2.03)

ADVERSE EVENTS:
Time Frame: Baseline to 6 months
Arm/Group | R-CAT | CAT Cognitive Adaptation Training
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/21
Other Adverse Events (participants affected / at risk) | 0/35 | 0/21

LIMITATIONS AND CAVEATS:
Not a a randomized trial. Due to the pandemic we were unable to compare groups choosing R-CAT/CAT versus those randomized. We did not get our desired number of participants. Also, some CAT in person treatment had to be conducted outside due to pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT04526067/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT04526067/ICF_000.pdf